CLINICAL TRIAL: NCT04344093
Title: Validation of a Connected Patch, an Alternative to Conventional Monitoring
Acronym: Patch
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019/11
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Anesthesia

STUDY DESIGN:
Intervention Model Description: Connected patch validation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Connected patch validation (Experimental)
  Interventions: Device: Patch validation

INTERVENTIONS:
Device: Patch validation — Use of connected patch to collect blood pressure, heart rate, respiratory rate, arterial oxygen saturation and temperature

SUMMARY:
The hypothesis is that this connected patch could be used in surgical departments to detect early a cardiovascular or respiratory complication and therefore to treat it without delay. However, it has not been validated in a hospital setting; that is the purpose of this project. This step of validating the connected monitoring object is required in different places: post-interventional surveillance room that approaches a conventional hospital room, and operating room where artifacts are numerous. Validation will be done by comparing data from General Electric's conventional monitors, with data from patches.

DETAILED DESCRIPTION:
When patients operated on outside intensive care or intensive care units are hospitalized, vital signs are collected intermittently by various conventional devices. During the follow-up period of these patients, it is possible that abnormal vital signs that may identify clinical deterioration may appear a few minutes to a few hours before a serious adverse event (infection etc.) occurs. These signals often go unnoticed due to infrequent monitoring.

The establishment of teams to ensure a rapid response would improve the safety of hospitalized patients for whom the detection of abnormal vital signs predictive of clinical deterioration would generate an alarm. This system is based on the identification of patients at risk and the rapid intervention of the team.

One of the crucial issues is therefore the speed of the alarm and its reliability.

The evolution of electronic technology offers the possibility of using inexpensive portable devices (connected patches) that can provide information on vital signs in real time. Vital signs collected by these devices could be analyzed to predict clinical deterioration prior to hospital staff visits, especially at night and on weekends when staffing levels are generally lower.

The connected patch used in this research is the Devinnova company's device "myAngel VitalSigns". The long-term objective would be to be able to use this connected patch in surgical departments to detect early a complication, particularly of a cardiovascular or respiratory nature, and therefore to treat it without wasting time. However, it has not been validated in a hospital setting; that is the purpose of the project.

The objective of this research is therefore to validate Devinnova's connected patch in different locations: post-interventional surveillance room that approaches a conventional hospital room, operating room where artifacts are numerous.

ELIGIBILITY:
Inclusion Criteria:

* patient over 18 and under 85 years of age
* patient requiring general anesthesia for extra-thoracic surgery
* the patient's position during the operation is in supine position only
* patient affiliated to or benefiting from social security, excluding State Medical Assistance
* patient with written consent

Exclusion Criteria:

* pregnant or breastfeeding patients
* patients known to have severe skin reactions to adhésives
* patient whose surgical procedure prevents the patch from being placed (intervention on the thorax)
* patients deprived of their liberty or under guardianship

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2022-05-29 (Estimated); Study Completion 2022-06-03 (Estimated)

PRIMARY OUTCOMES:
Concordance of blood pressure value measured by 2 different devices during the postoperative stay in the post-operative period in the post-anesthesia care unit | 36 hours maximum after the surgery
  Comparison between blood pressure measured by conventional medical monitoring device and by connected patch
Concordance of heart rate value measured by 2 different devices during the postoperative stay in the post-operative period in the post-anesthesia care unit | 36 hours maximum after the surgery
  Comparison between heart rate measured by conventional medical monitoring device and by connected patch
Concordance of respiratory rate value measured by 2 different during the postoperative stay in the post-operative period in the post-anesthesia care unit | 36 hours maximum after the surgery
  Comparison between respiratory rate measured by conventional medical monitoring device and by connected patch
Concordance of arterial oxygen saturation value measured by 2 different devices during the postoperative stay in the post-operative period in the post-anesthesia | 36 hours maximum after the surgery
  Comparison between arterial oxygen saturation measured by conventional medical monitoring device and by connected patch
Concordance of temperature value measured by 2 different devices during the postoperative stay in the post-operative period in the post-anesthesia care unit | 36 hours maximum after the surgery
  Comparison between temperature measured by conventional medical monitoring device and by connected patch

SECONDARY OUTCOMES:
Concordance of blood pressure value measured by 2 different devices during anesthesia | During anesthesia
  Comparison between blood pressure measured by conventional medical monitoring device and by connected patch
Concordance of heart rate value measured by 2 different devices during anesthesia | During anesthesia
  Comparison between heart rate measured by conventional medical monitoring device and by connected patch
Concordance of respiratory rate value measured by 2 different devices during anesthesia | During anesthesia
  Comparison between respiratory rate measured by conventional medical monitoring device and by connected patch
Concordance of arterial oxygen saturation value measured by 2 different devices during anesthesia | During anesthesia
  Comparison between arterial oxygen saturation measured by conventional medical monitoring device and by connected patch
Concordance of temperature value measured by 2 different devices during anesthesia | During anesthesia
  Comparison between temperature value measured by conventional medical monitoring device and by connected patch
Blood pressure artifact | From beginning of anesthesia to 36 hours
  An artifact is defined as any value that deviates from a physiologically plausible range or by a deviation > 50% from the previous value unless this value is followed by a value equal to ± 25%
Heart rate artifact | From beginning of anesthesia to 36 hours maximum after the surgery
  An artifact is defined as any value that deviates from a physiologically plausible range or by a deviation > 50% from the previous value unless this value is followed by a value equal to ± 25%
Respiratory rate artifact | From beginning of anesthesia to 36 hours maximum after the surgery
  An artifact is defined as any value that deviates from a physiologically plausible range or by a deviation > 50% from the previous value unless this value is followed by a value equal to ± 25%
Arterial oxygen saturation artifact | From beginning of anesthesia to 36 hours maximum after the surgery
  An artifact is defined as any value that deviates from a physiologically plausible range or by a deviation > 50% from the previous value unless this value is followed by a value equal to ± 25%
Acceptability of connected patch | During the surgery and 36 hours maximum after the surgery
  The patient will be asked to evaluate its acceptance of the sensor using a 4-point Likert scale (from 0 = intolerable to 4 = no problem at all)

CONTACTS AND LOCATIONS:
Overall Officials: Marc FISCHLER, MD, Study Chair — Hopital Foch
Locations (1):
- Hopital FOCH, Suresnes, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be available in the Dryad repository
Supporting Information: Analytic Code
Time Frame: After publication in a peer-review journal .No limit in time
Access Criteria: No criteria
URL: https://datadryad.org/stash

REFERENCES:
- [Derived] Le Guen M, Squara P, Ma S, Adjavon S, Trillat B, Merzoug M, Aegerter P, Fischler M. Patch validation: an observational study protocol for the evaluation of a multisignal wearable sensor in patients during anaesthesia and in the postanaesthesia care unit. BMJ Open. 2020 Sep 25;10(9):e040453. doi: 10.1136/bmjopen-2020-040453. PMID 32978206